CLINICAL TRIAL: NCT00717249
Title: Vistakon Investigational Contact Lenses Worn for Daily Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR-1513
Record Dates: First submitted 2008-07-15; First posted 2008-07-17 (Estimated); Results first posted 2016-05-26 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test Lens (Experimental): galyfilcon A contact lens with a silver additive
  Interventions: Device: galyfilcon A with a silver additive
- Control Lens (Active Comparator): galyfilcon A control contact lens
  Interventions: Device: galyifilcon A control lens

INTERVENTIONS:
Device: galyifilcon A control lens — Marketed daily wear contact lens
  Other Names: ACUVUE Advance with Hydraclear
  Arms: Control Lens
Device: galyfilcon A with a silver additive — Investigational daily wear contact lens
  Arms: Test Lens

SUMMARY:
This study compares the performance of an investigational contact lens to a currently marketed lens.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be at least 18 years of age.
2. Both males and females may be enrolled.
3. The subject must read, understand, and sign for themselves the STATEMENT OF INFORMED CONSENT and be provided with a copy of the form.
4. The subject is able and willing to wear soft contact lenses on a daily basis for a six month duration.

Exclusion Criteria:

1. The subject must be free of Grade 2 or greater slit lamp findings (edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection, and other ocular abnormality), which would contraindicate contact lens wear.
2. Any active ocular (i.e. corneal infiltrates, conjunctiva, lids, and intraocular) infection or inflammation of an allergic, bacterial, or viral etiology.
3. Entropion, ectropion, chalazia, recurrent styes, glaucoma or glaucoma suspect, history of recurrent corneal erosions and aphakia.
4. The following medications are prohibited (at lease one week prior to enrollment): oral retinoid isoretinoin (e.g. Accutane), oral tetracyclines, topical scopolamine, oral (e.g. antihistamines (e.g. Seldane, Chlor-Trimeton, and Benadryl), and ophthalmic antihistamic Beta-adrenergic blockers (e.g. Propranolol, Timolol, and Practolol), systemic steroids, and and prescribed or OTC ocular medication. Any prescription or PTC medications or preparations containing silver.
5. Moderate or above corneal distortion by keratometry.
6. Known allergy to silver, silver ions, or silver containing compounds.
7. Abnormal discoloration of the cornea and/or conjunctiva.
8. Routine exposure to silver, silver ions, or silver containing compounds.
9. The subject must be free of systemic diseases which may interfere with contact lens wear: diabetes, hyperthyroidism, recurrent herpes simplex/zoster, Sjogren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases (e.g. AIDS)
10. Free of systemic and infectious diseases: hepatitis and tuberculosis.
11. Subjects must be HIV negative.
12. The subject must not be currently be pregnant or lactating (Subject becoming pregnant during the study will be discontinued).
13. The subject's eyes must be best corrected to a visual acuity of 20/30 or better in each eye.
14. The subject must not have more than 1.00D of refractive astigmatism in either eye.
15. The subject's distance spherical contact lens prescription must be between -1.00D and -6.00D.
16. The subject must not be monovision corrected.
17. The subject must have no history of solution reaction to Opti-free RepleniSH MPDS-No Rub Solution.
18. The subject must not have any previous history or signs of a contact lens related corneal inflammatory event (i.e. past peripheral ulcers or round peripheral scars)
19. The subject must not have participated in a device or pharmaceutical clinical trial within 30 days prior to study enrollment.
20. The subject must not have had an eye injury within 8 weeks prior to study enrollment.
21. The subject must not have had previous eye surgery.
22. The subject must be successfully trial fitted with the study contact lenses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 529 (Actual)
Dates: Start 2007-08; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Cole, Cole, and Krohn, Fresno, California
  - Dr. James R. Dugue Family Optometrist, Mission Viejo, California
  - Fukai and Associates, Louisville, Colorado
  - Baymeadows Vision Center, Jacksonville, Florida
  - Eyecare Associates, Bloomington, Illinois
  - Advantage Eyecare Associates, LLC, Neodesha, Kansas
  - InSight Eyecare, Warrensburg, Missouri
  - Spectrum Eyecare, Jamestown, New York
  - Drs. Quinn, Quinn and Associates, Athens, Ohio
  - Dr. Michael H. Greenburg, Inc., Chagrin Falls, Ohio
  - Central Ohio Eyecare, Columbus, Ohio
  - James W. Kershaw OD, Inc., North Olmsted, Ohio
  - West Hills Vision Center, Moon Township, Pennsylvania
  - Nittany Eye Associates, State College, Pennsylvania
  - Research Across America, Wyomissing, Pennsylvania
  - Dr. David W. Ferris and Associates, Warwick, Rhode Island
  - Premier Vision, Amarillo, Texas
  - William J. Bogus OD, Salt Lake City, Utah
  - The Eye Speciliasts, Ltd, Virginia Beach, Virginia
  - Snowy Range Vision Center, Laramie, Wyoming

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 529 subjects were enrolled in this study. Of those enrolled subjects, 33 did not meet the eligibility criteria and 496 were randomized to either the test or control lens using a 2:1 allocation. Of those randomized subjects 491 were successfully dispensed. Of the dispensed subjects 454 subjects completed the study.
Groups:
- Galyfilcon A w/ Silver; Galyfilcon A: Subjects that were randomized to receive the galyfilcon A contact lens with a silver additive during the entire course of the study.
Period: Overall Study
Arm/Group | Galyfilcon A w/ Silver | Galyfilcon A
Started | 326 | 165
Completed | 304 | 150
Not Completed | 22 | 15
Not completed — Lens Discomfort | 4 | 1
Not completed — Unsatisfactory visual Response | 0 | 2
Not completed — Adverse Event | 4 | 2
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Pregnancy | 6 | 3
Not completed — Protocol Violation | 0 | 2
Not completed — Subject became Ineligible | 1 | 1
Not completed — Unsatisfactory Physiological Response | 0 | 1
Not completed — Gastric Surgery | 0 | 1
Not completed — Diagnosed with Diabetes | 1 | 0
Not completed — Diagnosed with Multiple Scletosis | 1 | 0
Not completed — Subject relocated | 1 | 0
Not completed — Headaches | 1 | 0

BASELINE CHARACTERISTICS:
Population: All subjects that were dispensed a study lens.
Groups:
- Galyfilcon A: Subjects that were randomized to receive the galyfilcon A contact lens during the entire course of the study.
- Total: Total of all reporting groups
Arm/Group | Galyfilcon A w/ Silver | Galyfilcon A | Total
Number analyzed (Participants) | 326 | 165 | 491
Age, Continuous [Mean (Full Range); unit: years] | 31.9 [18 to 60] | 29.8 [18 to 51] | 30.9 [18 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 226 | 98 | 324
  Male | 100 | 67 | 167
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 5 | 4 | 9
  White | 304 | 147 | 451
  African American | 5 | 3 | 8
  Native American | 0 | 1 | 1
  Asian - Indian | 2 | 0 | 2
  Hispanic | 8 | 9 | 17
  Other | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 326 | 165 | 491

OUTCOME MEASURES:

1. Primary Outcome: Slit Lamp Findings
Description: Each subjects' eye was examined using a bio-microscope. Slit lamp findings were graded using a 5- point scale. (Grade 0, 1, 2, 3 and 4). The data was dichotomized by creating 2 groups. Eyes with Grade 3 or Grade 4; eyes with Grade 2 or lower. The number of eyes with Grade 3 or Grade 4 was reported.
Time Frame: 6 months
Population: The analysis population consists of subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: Number of Subject Eyes
Units Other Than Participants: Subject Eyes
Arm/Group | Galyfilcon A w/ Silver | Galyfilcon A
Number analyzed (Participants) | 304 | 150
Number analyzed (Subject Eyes) | 608 | 300
Number of Subject Eyes | 7 | 2

2. Primary Outcome: Subject Reported Symptoms
Description: Subjects were asked "Have you experienced any symptoms or problems since your last visit?" at each visit and responded 'yes' or 'no' for each eye; at each visit(baseline, 2-, 4-, 12- and 26- week follow-up evaluations). If a subject responded 'yes' then the symptoms was classified into one of the four categories, "Dryness", "Other", "Cloudy/ Blurry / Hazy", "Irritation / Discomfort". The percentage of each response across all visits was reported.
Time Frame: 6 months
Population: The analysis population consists of subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: Percentage of Observations
Units Other Than Participants: Number of Observations
Arm/Group | Galyfilcon A w/ Silver | Galyfilcon A
Number analyzed (Participants) | 304 | 150
Number analyzed (Number of Observations) | 2548 | 1260
Percentage of Observations
  Dryness | 9.9 | 6.3
  Other | 4.9 | 4.0
  Cloudy/ Blurry / Hazy | 2.8 | 2.5
  Irritation / Discomfort | 2.8 | 2.3

3. Primary Outcome: Visual Acuity
Description: Binocular LogMAR Visual Acuity was taken under low luminance and high contrast conditions using ETDRS acuity charts.
Time Frame: 6 months
Population: The analysis population consists of subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Galyfilcon A w/ Silver | Galyfilcon A
Number analyzed (Participants) | 304 | 150
LogMAR | 0.004 (0.0891) | -0.009 (0.0866)

4. Primary Outcome: Average Contact Lens Wear Time
Description: The Contact lens wear time for the study contact lenses was collected for each subject. The average wear time for each contact lens was reported.
Time Frame: 6 Months
Population: The analysis population consists of subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Full Range); unit: time in hours
Arm/Group | Galyfilcon A w/ Silver | Galyfilcon A
Number analyzed (Participants) | 304 | 150
time in hours | 14.0 [13.92 to 14.03] | 14.0 [13.95 to 14.04]

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 6 months.
Arm/Group | Galyfilcon A w/ Silver | Galyfilcon A
Serious Adverse Events (participants affected / at risk) | 0/326 | 1/165
Other Adverse Events (participants affected / at risk) | 0/326 | 0/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galyfilcon A w/ Silver (N=326) | Galyfilcon A (N=165)
Iritis (Eye disorders) | 0 (0) | 1 (1) — Note from Dr. Not Lens Related. Possible Cause: "Iritis secondary to cornea culture"

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days